CLINICAL TRIAL: NCT05400148
Title: Dose and Concentration Relationship of Bupivacaine for Pericapsular Nerve Group Block in Hip Surgery
Brief Title: Dose and Concentration Relationship for PENG Block in Hip Surgery
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Onur Okur, Principal Investigator, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 108
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Hip Fractures; Post Operative Pain
Keywords: hip fracture; peripheral nerve blocks; postoperative pain; bupivacaine volume
MeSH Terms: conditions — Hip Fractures; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- low volume: This cohort will include the patients to whom an analgesic PENG block was administered with a bupivacaine solution volume of up to 20 ml in a dose of 2.5mg/kg-1. This cohort is anticipated to have 56 participants.
  Interventions: Drug: Bupivacaine Hydrochloride
- high volume: This cohort will include the patients to whom an analgesic PENG block was administered with a bupivacaine solution volume more than 20 ml in a dose of 2.5mg/kg-1. This cohort is anticipated to have 56 participants.
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — Patients who were administered an analgesic PENG block with a dose of 2.5mg/kg with either lov (<20ml) or high volume (>20ml)
  Other Names: PENG block

SUMMARY:
A number of peripheral nerve blocks are routinely performed in patients who will undergo orthopedic hip surgery for pain relief. Proximal extensor group nerve (PENG) block is one such field block which is used for this purpose and could be performed both before and after the operation. When used before surgery, PENG block is reported to be beneficial in alleviating pain during positioning for spinal anesthesia. Furthermore, some studies suggest a high volume block may increase the analgesic effect of the block. In this perspective, this study aims to observe the effects of different volumes of local anesthetic (bupivacaine) at the same dose used for PENG block in hip fracture positioning for spinal anesthesia.

The investigator hypothesizes that a high volume (>20ml) PENG block will reduce pain during positioning compared to a low volume PENG block.

DETAILED DESCRIPTION:
This prospective observational study will be conducted between 04.07.2022-04.01.2023 in the orthopedic operating rooms of T.C. Ministry of Health University of Health Sciences Prof. Dr. Cemil Taşçıoğlu City Hospital. Patients over the age of 18 who are scheduled for hip fracture under spinal anesthesia meeting the inclusion criteria and who agree to participate in the study by signing a consent form will be included. Patients will be surveyed about the amount of pain they suffer with numerical rating scale (NRS) four times; firstly, 15 minutes after the block at rest, then, a second time with a 10 degree hip flexion, after that a third time when patient is given sitting position for spinal anesthesia, and lastly, 24 hours after the surgery. Age, height, weight, gender, co-morbidities, American Society of Anesthesiologists physical condition (ASA) scores, time of block administration, whether an intraoperative complication developed (hypotension, tachycardia, bradycardia, inotropic need, desaturation), local anesthetic (bupivacaine) volume used for PENG block will be recorded from the anesthesia charts. Twenty-four hours after the surgery patients will be questioned for nausea, vomiting and urinary retention. At this point the 4 A's test (4AT) will be performed to detect any presence of delirium. Postoperative iv analgesic treatments and mobilization times(if mobilized) of the patients will be recorded from patient charts. Resulting data for low volume (less than or equal to 20ml) and high volume PENG blocks will be compared.

It is expected that a total of 112 patients will be recruited for this study. A power analysis revealed that it is necessary to recruit at least 102 patients, when effect size d is assumed to be 0.5 ( for medium difference) for a 0.05 alpha error with a %80 power. Taking in account a 10% follow-up loss we planned to recruit 112 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who consent to participate and;
* Patients who are scheduled for hip surgery under spinal anaesthesia,
* Patients who have no neurocognitive disorders that impair cooperation and communication (e.g Alzheimer's disease, Parkinson's disease, senile dementia),
* Patients who have no local anaesthetic allergies,
* Patients to whom an analgesic PENG block was administered preoperatively to facilitate sitting position during spinal anaesthesia will be included.

Exclusion Criteria:

* Patients under the age of 18,
* Patients who decline to participate,
* Patients who are scheduled for hip surgery under general anaesthesia
* Patients who have neurocognitive disorders
* Patients who have local anaesthetic allergies
* Patients to whom an analgesic PENG block was NOT administered preoperatively to facilitate sitting position during spinal anaesthesia will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected consecutively from those who are admitted to a tertiary care center with a diagnosis of hip fracture and scheduled for a hip surgery in a tertiary care center, until the required sample size is achieved.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Sitting pain | 30 minutes after PENG block is performed
  Pain score according to numerical rating scale when patient is brought to sitting position for spinal anesthesia. Numeric rating scale is a patient's self reported pain score between a minimum of "0" and a maximum of "10". Higher numbers indicate worse pain. A score of "0" means that patient suffers no pain at all while a score of "10" means they suffer the worst pain possible.

SECONDARY OUTCOMES:
Block pain at rest | 15 minutes after PENG block is performed
  Pain score at rest according to numerical rating scale after PENG blok is performed. Numeric rating scale is a patient's self reported pain score between a minimum of "0" and a maximum of "10". Higher numbers indicate worse pain. A score of "0" means that patient suffers no pain at all while a score of "10" means they suffer the worst pain possible.
Block pain with movement | 15 minutes after PENG block is performed
  Pain score with 10 degree flexion according to numerical rating scale after PENG. Numeric rating scale is a patient's self reported pain score between a minimum of "0" and a maximum of "10". Higher numbers indicate worse pain. A score of "0" means that patient suffers no pain at all while a score of "10" means they suffer the worst pain possible.
Postoperative pain | Postoperative 24th hour
  Pain score at rest according to numerical rating scale postoperatively. Numeric rating scale is a patient's self reported pain score between a minimum of "0" and a maximum of "10". Numbers increase with increasing pain and a score of "0" means that patient suffers no pain at all and "10" means they suffer the worst pain possible.
Breakthrough analgesic use | Postoperative 24th hour
  Existence and amount of breakthrough analgesics used
Delirium | Postoperative 24th hour
  Existence of delirium according to 4AT score

CONTACTS AND LOCATIONS:
Overall Officials: Onur OKUR, Principal Investigator — Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Locations (1):
- Prof. Dr. Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)